CLINICAL TRIAL: NCT03400826
Title: A Double-blinded, Phase II, Randomized Control Trial to Study the Effects of Simvastatin in Patients With Uterine Leiomyoma
Brief Title: Effects of Simvastatin on Uterine Leiomyoma Size
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00149869; 1R01HD094380-01 (NIH)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Fibroid Uterus; Fibroid Tumor; Leiomyoma; Fibromyoma; Leiomyoma, Uterine
Keywords: simvastatin; fibroids; medical management; uterine fibroids; leiomyoma
MeSH Terms: conditions — Leiomyoma | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The 30 participants randomized in this group will intake Simvastatin 40mg / day of orally at the same time in the evening, every day for the study duration of 12 weeks prior to undergoing hysterectomy/ myomectomy. The fibroid samples will be collected after the surgery to evaluate the effects of the study medication on the fibroid tissue.
  Interventions: Drug: Simvastatin 40mg
- Placebo Group (Placebo Comparator): The 30 participants randomized in this group will intake Placebo 40mg / day orally at the same time in the evening every day for the study duration of 12 weeks prior to undergoing hysterectomy/ myomectomy. The fibroid samples will be collected after the surgery to evaluate the effects of the study medication on the fibroid tissue.
  Interventions: Drug: Placebo 40 mg

INTERVENTIONS:
Drug: Simvastatin 40mg — The Treatment Group subjects will orally intake encapsulated Simvastatin 40 mg tablets daily for the 12 weeks duration with water in the evening.
  Other Names: Simvastatin
  Arms: Treatment Group
Drug: Placebo 40 mg — The Placebo group will orally intake encapsulated Starch 1500, 40 mg Placebo for 12 weeks duration with water in the evening.
  Other Names: Starch 1500 encapsulated
  Arms: Placebo Group

SUMMARY:
The study aims to study the effect of simvastatin on the size of uterine fibroids.

DETAILED DESCRIPTION:
The study is a phase II double blinded clinical trial to determine feasibility, safety and preliminary clinical efficacy of simvastatin to reduce leiomyoma size. Women with symptomatic fibroids planned to undergo surgical management for fibroids such as hysterectomy or myomectomy will be screened for participation. The eligible women will undergo pre-study evaluation to ascertain study eligibility.The study will enroll 60 participants in total, half will receive simvastatin and the other half will receive a placebo. The study drug and placebo will be an add on to the participants ongoing medical management of fibroids until surgery. The participants will be monitored at intervals for the effect of the drug on fibroid size and symptoms using ultrasound and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed written consent.
* Gender: female.
* Age: 18-55 years at time of signing consent.
* BMI of subjects: < 45 kg/m2.
* Uterine fibroids:
* Diagnosed by ultrasound (MRI will be used only if ultrasound is inconclusive).
* Number: any number of fibroids.
* Location: submucosal or intramural.
* At least one fibroid of diameter > 3cm.
* Symptoms: one or more of the following symptoms of heavy menstrual bleeding (HMB), defined as: Experienced cyclic (22 to 35 days) abnormal uterine bleeding (heavy or prolonged) in at least 3 of the last 6 menstrual periods, including menstrual bleeding lasting 5 or more days or heavy bleeding per participant recall. Examples of heavy bleeding may include, but are not limited to the following:
* Requires the use of double protection to manage menstrual bleeding.
* Menstrual bleeding accompanied by the sensation of "gushing" or "flooding".
* Saturates more than 1 tampon or sanitary pad per hour for 3 or more consecutive hours.
* Regularly needs to change the tampon or sanitary pad at night or regularly soils bedclothes.
* Heavy bleeding that affects work, school, or social activities.
* Pelvic pain/ pressure likely caused by fibroids.
* Plan for surgery (hysterectomy or myomectomy).
* Normal Pap smear within the last year.
* Use of contraception during study such as non-hormonal oral contraceptives, intrauterine devices (IUD)/ intrauterine systems (IUS), barrier contraceptives, abstinence or sterilization.

Exclusion Criteria:

* Pregnancy or lactation.
* Previous or current uterine, cervical or ovarian cancer.
* Current endometrial hyperplasia or history of atypical endometrial hyperplasia. Endometrial biopsy will be done during screening (if not done within last 12 months).
* Suspicion of leiomyosarcoma.
* Recent rapid growth of fibroids (i.e. doubling in size within 1-6 months period).
* Unevaluated gynecologic abnormalities (unexplained vaginal bleeding, cervical dysplasia, or abnormal adnexal/ovarian mass).
* Menopausal status.
* Surgery is urgently indicated (< 3 months) for medical or social reasons.
* Hemoglobin ≤ 6 g/dL.
* Currently enrolled in another investigational study.
* Mental condition or other barrier preventing informed written consent.
* Allergy or hypersensitivity to simvastatin.
* Current use of simvastatin or other drugs of the same class.
* Concomitant administration of strong CYP3A4 inhibitors including itraconazole, ketoconazole, posaconazole, voriconazole, erythromycin, clarithromycin, telithromycin, HIV protease inhibitors, boceprevir, telaprevir, nefazodone, and cobicistat-containing products.
* Concomitant administration of gemfibrozil, cyclosporine, or danazol, verapamil, diltiazem, amiodarone, diltiazem, dronedarone, amlodipine, ranolazine, lomitapide, and grapefruit juice.
* Active liver disease, which may include unexplained persistent elevations in hepatic transaminase levels.( elevation of aspartate transaminase and/or alanine transaminase > 2 s.d. above the normal range at screening visit)
* Known increased risk or diagnosis of a myopathy.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Tumor size volume pre and post study intervention | Change from baseline to 12 weeks post intervention
  Tumor size measured by ultrasound imaging comparing tumor volume using ultrasound imaging. The volume will be reported in Centimeter cubes. The largest radius of the tumor will be used to calculate the volume, this will be measured in centimeters.

SECONDARY OUTCOMES:
Clinical symptom improvement as determined by the Uterine Fibroid Symptom and Health Related Quality of Life Questionnaire. | At visit 1 (Screening), At visit 2 (start of the study drug intake), visit 3 (6 weeks after start of the study drug), visit 4( 12 weeks after start of the study drug), and follow up visit at 2 and 6 weeks post hysterectomy
  The questionnaire used is the Uterine Fibroid Symptom and Health Related Quality of Life Questionnaire. This questionnaire is an effective and validated tool for detecting differences in symptom severity and health-related quality of life among patients with uterine fibroids. The scale for this questionnaire denotes symptom severity with lowest and highest possible scores of 8 and 40 respectively. Higher scores indicate greater severity of symptoms.
Adherence to the recommended treatment dosing | At Visit 3 (6 weeks after start of study drug), and Visit 4 (12 weeks after start of the study drug)
  Based on review of patient diaries and counting of left over medications bought back by the subject. This will be reported as an overall percentage.
Subject retention | At visit 2 (start of the study drug intake), visit 3 (6 weeks after start of the study drug), visit 4 (12 weeks after start of the study drug), and follow up visit at 2 and 6 weeks post hysterectomy.
  Based on presence at follow up visits to the study site. This will be determined as a simple percentage of subjects that stay in the study until the last visit.

OTHER OUTCOMES:
Adverse events reporting by organ systems | At visit 2 (start of the study drug intake), visit 3 (6 weeks after start of the study drug), visit 4 (12 weeks after start of the study drug), and follow up visit at 2 and 6 weeks post hysterectomy.
  Based on patient reporting and study team evaluation utilizing CTCAE v.4

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Borahay, MD, PhD, Principal Investigator — Johsn Hopkins School Of Medicine
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No